CLINICAL TRIAL: NCT05596630
Title: A Single-center, Unblinded, Single-arm, Prospective Trial of Stereotactic Body Radiation Therapy for the Safety and Prognosis of Small Intrahepatic Recurrent Hepatocellular Carcinoma
Brief Title: Stereotactic Body Radiation Therapy for the Safety and Prognosis of Small Intrahepatic Recurrent HCC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-0771
Record Dates: First submitted 2022-10-25; First posted 2022-10-27 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-01

CONDITIONS: Carcinoma; Hepatocellular
Keywords: Stereotactic Body Radiation Therapy; Recurrent Hepatocellular Carcinoma; Small liver cancer
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Stereotactic body radiation therapy (Experimental): Radiation dose: Greater than or equal to 40Gy/4-5F, complete treatment within 1 week.
  Interventions: Radiation: Stereotactic body radiation therapy

INTERVENTIONS:
Radiation: Stereotactic body radiation therapy — Stereotactic body radiotherapy for small intrahepatic recurrent HCC. Radiation dose: Greater than or equal to 40Gy/4-5F, complete treatment within 1 week.

SUMMARY:
Primary liver cancer is one of the common malignant tumors in China, of which hepatocellular carcinoma (HCC) accounts for 85%-90%. It is worth noting that the recurrence rate of liver cancer is greater than 10% at 1 year after surgery, while the recurrence rate in 5 years reaches 70-80%.

Stereotactic body radiation therapy (SBRT) refers to a kind of radiotherapy technology to achieve a steep dose gradient and achieve high-precision position and high-dose fractionated irradiation. The rapid dose drop-down enables SBRT to maximize the protection of normal tissues around the tumor, and it often requires only 1-5 times of high-dose fractionated irradiation to complete the course of treatment.SBRT may play an important role in the treatment of small intrahepatic recurrence HCC, but there is still a lack of evidence of high-level prospective studies.

We intend to conduct a single-center, prospective, clinical study to further elaborate the efficacy and safety of SBRT in the treatment of small intrahepatic recurrent HCC.

DETAILED DESCRIPTION:
Patients with recurrent small hepatocellular carcinoma after surgery or local ablation therapy are chosen for this study. A total of 40 patients will be scheduled to be enrolled. The patients enrolled will be treated with SBRT with no adjuvant therapy, and they will be followed up according to the plan.

ELIGIBILITY:
Inclusion Criteria:

* 1. Clinical or pathological diagnosis of HCC without lymph node and distant metastasis.

  2. Previous surgery or radiofrequency ablation, no recurrence within 6 months. 3. Early stage liver cancer within Milan criteria : (1) single tumor diameter less than 5 cm; (2) not more than three foci of tumor, each one not exceeding 3 cm; (3) no angioinvasion; (4) no extrahepatic involvement.

  4. The remnant liver volume beyond the radiotherapy target area should be greater than 700ml.

  5. No serious hematological, heart, lung, hepatic, renal dysfunction and immunodeficiency.

  6. Hemoglobin (Hb)≥8g/dL ; white blood cell (WBC) ≥ 2*10^9/L ; neutrophils (ANC) ≥ 1.0* 10^9/L ; platelet (Pt) ≥ 50*10^9/L.

  7. Men or women with fertility are willing to take contraceptive measures in the trial.

  8. ECOG score standard 0 ~ 1 ; child-pugh score A-B . 9. Expected survival period > 3 months. 10. Voluntary participation and signing of informed consent.

Exclusion Criteria:

* 1. Patients who have undergone antitumor therapy for liver cancer. 2. Obvious cirrhosis, recent hematemesis due to portal hypertension, Child-Pugh score ≥10 points.

  3. Total bilirubin exceed the upper limit of normal 1.5 times, aspartate aminotransferase (ALT), alanine aminotransferase (AST) exceed the upper limit of normal 2.5 times, ICGR15≥40%.

  4. Patients undergoing major surgery within 1 month of study initiation. 5. Patients with previous history of malignancy (excludes tumor-free survival after treatment of basal cell carcinoma of the skin and carcinoma of the cervix in situ for more than 3 years).

  6. Participants in other clinical trials within 30 days prior to study treatment.

  7. The distance between the tumor and the gastrointestinal tract < 0.5 cm. 8. Pregnancy, lactation or those with fertility but without contraceptive measures.

  9. Patients with drug addiction such as drugs, long-term alcoholism, and AIDS. 10. Patients have an uncontrollable epileptic seizure, or lose insight due to mental illness.

  11. Patients with severe allergic history or specific constitution. 12. Researchers consider it inappropriate to participate in the test.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Local control rate（LC） | up to 24 months after SBRT
  The treatment efficacy is assessed by calculation of local control rate of irradiated locations according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 criteria (complete response + partial response + stable disease)

SECONDARY OUTCOMES:
Short time Safety profile of SBRT | up to 3 months after SBRT
  Toxicities appeared during SBRT treatment and up to 3 months after SBRT. Toxicities will be assessed by the evaluation of intensity and incidence of the Adverse Events (AE) displayed by patients. The intensity of each AE will be classified according to Common Terminology Criteria for Adverse Events (CTCAE) version 4.0
Overall response rate (ORR) | up to 24 months after SBRT
  According to RECIST v1.1, the proportion of patients with at least one complete response (CR) or partial response (PR) (%)
Overall survival (OS) | up to 24 months
  The time between the date of SBRT and death from any cause
Local recurrence rate (LRR) | up to 24 months after SBRT
  Rate of intrahepatic hepatocellular carcinoma recurrence
Progression-free survival (PFS) | up to 24 months
  The time between the date of SBRT and the date of radiographic progression as defined by RECIST1.1

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No